CLINICAL TRIAL: NCT06646497
Title: Evaluation of an Optimized Allogeneic Hematopoietic Stem Cell Transplantation Protocol With Post-transplant Cyclophosphamide in Patients Aged 40 to 60 Years Old With Acquired Aplastic Anemia Refractory or in Relapse After Immunosuppression
Brief Title: Indication of HSCT in Patients With Refractory/Relapse AA After First-line Standard Immunosuppressive Therapy Aged More Than 40 Years
Acronym: APARR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230832
Record Dates: First submitted 2024-09-13; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-08

CONDITIONS: Aplastic Anemia
Keywords: Refractory/relapse idiopathic anemia; Idiopathic aplastic anemia; Hematopoietic stem cell transplantation; Post-transplantation cyclophosphamide
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Intervention Model Description: A phase II multicenter, national, prospective, single-arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allogeneic hematopoietic stem cell transplantation Stem cell source only Bone Marrow (Experimental)
  Interventions: Biological: Allogeneic hematopoietic stem cell transplantation Stem cell source only Bone Marrow

INTERVENTIONS:
Biological: Allogeneic hematopoietic stem cell transplantation Stem cell source only Bone Marrow — 1. Conditioning regimen Thymoglobulin (0.5/mg/kg à D-9, 2 mg /kg at D-8 and 2.5 mg/kg à D-7), Fludarabine (30mg/m2/day i.v: day -6 to day -2), pre-transplant, Cyclophosphamide (14.5 mg/kg/day i.v: day -6 and day -5), and Total Body Irradiation (2 Gray on day -1).
  2. Stem cell source Bone Marrow only. Target of 4 × 10^8 nucleated cells/kg recipient body weight. Granulocyte colony stimulating factor is given subcutaneously starting on day +5 at 5 mg/ kg/day until the absolute neutrophil count is greater than 1.5 × 10^9/L for 3 days.
  3. GVHD prophylaxis Cyclophosphamide 50 mg/Kg/day at D+3 and D+4. Tacrolimus (0,2 à 0,3 mg/kg/day per os divided into 2 doses or 0.05 to 0.1 mg/kg/d IVSE) and mycophenolate (MMF) will begin from D+5. In absence of GvHD, MMF will be stopped between D35 and D45 and Tacrolimus at day 365.
  4. Prevention of EBV reactivation Rituximab 150mg/m2 intravenously at Day+5 post HSCT (except patients and their donor with EBV serology and EBV PCR negative).

SUMMARY:
Outcomes for adult patients with Severe Aplastic Anemia (SAA) aged more than 40 years who are refractory or in relapse after first-line IST remain poor. Hematopoietic stem cell transplantation (HSCT) is the unic valid therapeutic option but results have always been disappointing in patients aged 40 years or older. The first cause of death after HSCT in those refractory/relapse SAA patients is still graft versus host disease (GvHD). Recently, new strategies to prevent GvHD, including T-cell replete grafts with administration of post-transplantation cyclophosphamide (PTCy), have revolutionized the field, notably in haplo-identical donor setting. Using marrow as source of stem cells and a PTCy strategy not only in haplo-identical donor setting but also in case of an available matched sibling or unrelated donor might prevent drastically GvHD and eventually be practice changing. Evaluating this new strategy is the main objectives of "APARR".

ELIGIBILITY:
Inclusion Criteria:

* Aged from 40 to 60 years old
* Suffering from acquired refractory severe idiopathic aplastic anemia after at least 6 months treatment with anti-thymocyte globulin, cyclosporine with Eltrombopag or in relapse
* Allograft validated in the National Multidisciplinary expertise meetings of the French reference centre for aplastic anemia
* With an available geno-identical donor or 10/10 matched donor or haploidentical donor
* With the absence of donor specific antibody detected in the patient with a MFI < 1500 (antibodies to the distinct haplotype between donor and recipient)
* Usual criteria for HSCT:

  * ECOG ≤ 2
  * No severe and uncontrolled infection
  * Cardiac function compatible with high dose of cyclophosphamide
  * With an adequate organ function ASAT and ALAT ≤ 3N, conjugated bilirubin ≤ 2N (or total bilirubin ≤ 2N if not available), clearance creatinine ≥ 50ml / min
* With health insurance coverage
* Women of childbearing potential and men must use contraceptive methods during their participation to the research and for 12 months and 6 months after the last dose of cyclophosphamide, respectively.
* Having signed a written informed consent

NB: The authorized contraceptive methods are: For women of childbearing age and in absence of permanent sterilization:

* oral, intravaginal or transdermal combined hormonal contraception,
* oral, injectable or transdermal progestogen-only hormonal contraception,
* intrauterine hormonal-releasing system (IUS),
* sexual abstinence (need to be evaluated in relation to the duration of clinical trial and the preferred and usual lifestyle of the participants).

For men in absence of permanent sterilization: sexual abstinence, condoms.

Individuals must meet all of the inclusion criteria as verified at the screening / inclusion visit to be eligible to participate at the study.

Exclusion Criteria:

Patients:

* With morphologic evidence of clonal evolution (patients with isolated bone marrow cytogenetic abnormalities are also eligible excepted chromosome 7 abnormalities and complex karyotype).
* With seropositivity for HIV or HTLV-1-2 or active hepatitis B or C and associated hepatic cytolysis
* Cancer in the last 5 years (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix)
* Pregnant (βHCG positive) or breast-feeding
* Yellow fever vaccine and all others live virus vaccines within 2 months before transplantation and during the research
* With uncontrolled coronary insufficiency, recent myocardial infarction < 6-month, current manifestations of heart failure according to NYHA (II or more), ventricular ejection fraction <50%
* With renal failure with creatinine clearance <50ml /min
* Any contraindication mentioned in the SmPC and the Investigator's brochure of all medicinal products planned to be used in the trial including conditioning regimen, GVHD prophylaxis, prevention of EBV reactivation, infection prophylaxis
* Known allergy or intolerance to all medicinal products and/or excipients planned to be used in the trial including conditioning regimen, GVHD prophylaxis, prevention of EBV reactivation, infection prophylaxis, according to Investigator's brochure and SmPC.
* Who have any debilitating medical or psychiatric illness, which precludes understanding the inform consent as well as optimal treatment and follow-up
* Under legal protection (tutorship or curatorship)
* Under state medical aid
* Participation to another interventional trial on a medicinal product or cell therapy

Individuals meeting any of the exclusion criteria as verified at the screening / inclusion visit will be ineligible to participate at the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
GRFS (Graft Versus Host Disease (GvHD) and Relapse/rejection-Free Survival) | 2 years after transplantation
  GRFS is a composite right-censored endpoint, defined as the time from HSCT to the first of the following events:
  * primary graft failure, defined as the absence of engraftment from aplasia at day 60 after graft (D0) (i.e., persistence of neutrophils< 500 AND platelets < 20 Giga/L)
  * secondary graft failure, defined as the reoccurrence of aplasia after engraftment (defined as both occurrence of neutrophils< 500 for 3 days and platelets < 20 Giga/L for 7 consecutive days)
  * grade 3-4 acute GVHD, according to the MAGIC CONSORTIUM 2016
  * severe chronic GVHD, according to the NIH classification
  * death, whatever the cause

SECONDARY OUTCOMES:
Neutrophil engraftment | At day 100
  Neutrophils engraftment will be defined as first day of 3 consecutive days with neutrophils >0.5 G/L.
  With donor chimerism> 85% on the total blood.
Platelets engraftment | At day 100
  Platelets engraftment will be defined as first day of 7 consecutive days with platelets >20 G/L.
  With donor chimerism> 85% on the total blood.
Absolute number of neutrophils | At 1 month
Absolute number of neutrophils | At 3 months
Absolute number of neutrophils | At 6 months
Absolute number of neutrophils | At 12 months
Absolute number of neutrophils | At 24 months
Absolute number of neutrophils | At day of last platelet and red blood cell transfusions (up to 24 months)
Absolute number of platelets | At 1 month
Absolute number of platelets | At 3 months
Absolute number of platelets | At 6 months
Absolute number of platelets | At 12 months
Absolute number of platelets | At 24 months
Absolute number of platelets | At day of last platelet and red blood cell transfusions (up to 24 months)
Acute GvHD incidence grade 2-4 | At 3 months
Chronic GvHD incidence | At 24 months
Severe chronic GvHD | At 24 months
Secondary graft failure | At 12 months
Secondary graft failure | At 24 months
Severe infections | At 1 month
  CTCAE grade 3-4
Severe infections | At 3 months
  CTCAE grade 3-4
Severe infections | At 6 months
  CTCAE grade 3-4
Severe infections | At 12 months
  CTCAE grade 3-4
Severe infections | At 24 months
  CTCAE grade 3-4
Incidence of cardiac toxicities | At 12 months
Incidence of Epstein Barr Virus (EBV) infection | At 12 months
Incidence of CytoMegaloVirus (CMV) infection | At 12 months
Mortality | At 12 months
Mortality | At 24 months
Overall survival | At 12 months
Overall survival | At 24 months
Quality Of Life questionnaire | Before transplantation - at baseline day 0
  Quality of life will be evaluated using PedsQL questionnaire. Scores varies from 0 to100, with higher scores associated with better health-related quality of life
Quality Of Life questionnaire | At 6 months
  Quality of life will be evaluated using PedsQL questionnaire. Scores varies from 0 to100, with higher scores associated with better health-related quality of life
Quality Of Life questionnaire | At 12 months
  Quality of life will be evaluated using PedsQL questionnaire. Scores varies from 0 to100, with higher scores associated with better health-related quality of life
Quality Of Life questionnaire | At 24 months
  Quality of life will be evaluated using PedsQL questionnaire. Scores varies from 0 to100, with higher scores associated with better health-related quality of life
Chimerism | At 1 month
  Proportion of patients with a donor chimerism of 85% or more
Chimerism | At 3 months
  Proportion of patients with a donor chimerism of 85% or more
Chimerism | At 6 months
  Proportion of patients with a donor chimerism of 85% or more
Chimerism | At 12 months
  Proportion of patients with a donor chimerism of 85% or more
Chimerism | At 24 months
  Proportion of patients with a donor chimerism of 85% or more
Immune reconstitution | At 1 month
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL.
Immune reconstitution | At 3 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL.
Immune reconstitution | At 6 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL.
Immune reconstitution | At 12 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL.
Immune reconstitution | At 24 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, France